CLINICAL TRIAL: NCT01003912
Title: Treatment of Early Infantile-Onset Lysosomal Storage Diseases With Fetal Umbilical Cord Blood (UCB) Transplantation
Brief Title: Fetal Umbilical Cord Blood (UCB) Transplant for Lysosomal Storage Diseases
Acronym: IUHST-001
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Patients were consented to screening but none were enrolled and proceeded with transplant.
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: Aldagen (Industry)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010188
Record Dates: First submitted 2009-10-20; First posted 2009-10-29 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Lysosomal Storage Diseases; Inborn Errors of Metabolism
Keywords: Lysosomal Storage Diseases; Inborn Errors of Metabolism; Krabbe; Infantile metachromatic leukodystrophy disease; MLD; Tay Sachs; Sandhoff; GM2 gangliosidoses; Pelizaeus-Merzbacher disease; PMD
MeSH Terms: conditions — Lysosomal Storage Diseases; Metabolism, Inborn Errors; Gangliosidoses, GM2; Pelizaeus-Merzbacher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: ALD-601 — ALD-601 is manufactured by Aldagen from the 20% compartment of the selected umbilical cord blood unit within 24 hrs of planned injection. A dose of ALD-601 that delivers 1 x 105 - 2 x 106 cells/kg of estimated fetal weight at day - 1 is suspended in 300 microliters of dialysis media.

SUMMARY:
The purpose of this study is to determine if it is safe to administer unrelated umbilical cord blood to pregnant women in their first trimester of pregnancy with a fetus that has a known diagnosis of certain lysosomal storage diseases. These diseases are known to cause severe and irreversible neurological disability in early infancy and which are lethal in childhood.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety of first trimester fetal stem cell therapy using unrelated donor partially HLA-matched stem and progenitor cells derived from human umbilical cord blood for the treatment of selected lysosomal storage diseases that are known to cause severe and irreversible neurological disability in early infancy and which are lethal in childhood.

This study is designed as a prospective phase I open-label single center trial. It is designed to asses the safety and feasibility of administration of ALD-601 UCB cells to first trimester fetuses known to be affected with a lethal lysosomal storage disease. The sample size is 12 patients enrolled in cohorts of size 3. Safety measures will be monitored by an independent DSMC in each of the 4 cohorts prior to proceeding to the next cohort.

Biological parents being considered for therapy will have HLA testing, mutation analysis for disease status, and psychological counseling. Mothers will have ultrasounds for gestational age and chorion villus testing for mutation analysis for Krabbe, MLD, Tay Sachs, Sandhoff, or PMD (whichever appropriate). A crown-rump length will be determined the day before the scheduled transfer. The fetal weight will be calculated from formula: Y (kg) = (2.9026 x 10-1) (X 2.6528). The estimated fetal weight at that gestational age would be about 0.5 ounces or 14 grams. A suitably matched unrelated umbilical cord blood will be identified and the 20% portion will be manipulated for the isolation of ALD-601 cells. ALD-601 (ALDHbr) cells are isolated by high speed flow sorting on the FACSAria (BD Biosciences). Upon completion of the sort, ALD-601 UCB cells are counted, viability is determined, and the cellular composition of the sample is measured by analytical flow cytometry using fluorescence antibodies to lineage marker for T-cells, granulocytes, monocytes, and erythrocytes. The content of ALDHbr cells is also confirmed by analytical flow cytometry. A dose of 1 x 105 - 2 x 106 cells/kg of estimated fetal weight is suspended in 300 microliters of Cellgenix Stem Cell Medium (CellGenix, Inc.). Release criteria will allow a maximum of 5 x 104 T cells/kg. If the sorted sample contains greater than 5 x 104 T cells/kg it is re-sorted using the FACSAria and re-evaluated for cell number, viability, and cellular content. Sterility testing will include Bac-T/ALERT cultures, endotoxin measurement (LAL), and gram stain. After meeting criteria for product release, ALD-601 is transported at 2-8 degree C in a validated cooler to Duke and released to the Stem Cell Laboratory. Duke personnel will transport the cooler containing the ALD-601 product to the ultrasound suite, where the medical team will allow the ALD-601 to warm briefly to room temperature prior to injection. Under continuous ultrasound guidance, a 22-gauge X 5 inch procedure needle will be used to puncture the fetal peritoneal cavity. 100 microliters of sterile saline will be instilled to confirm intraperitoneal placement. The stem cell infusion will then be injected through the needle followed by the injection of 200 microliters (dead space of the needle: 60 microliters) to displace all cells from the dead space of the needle. An ultrasound will be performed 24 hours later to confirm fetal viability. A subsequent ultrasound will be undertaken at 18 weeks gestation to confirm viability, assess detailed fetal anatomy and adequate serial fetal growth.

ELIGIBILITY:
Inclusion Criteria:

* Fetus with known enzymatic and, if possible, mutation diagnosis of selected lysosomal storage diseases, and history of enzymatic or mutation diagnosis of a previously affected family member.
* Krabbe disease
* Infantile metachromatic leukodystrophy disease (MLD)
* Tay Sachs or Sandhoff (GM2 gangliosidoses) disease
* Pelizaeus-Merzbacher disease (PMD).
* Both parents have the "at risk" genotype
* Both parents agree to psychological counseling prior to CVS
* Both parents agree to delivery of subject at Duke University
* Gestational age of < 9 weeks by sure menstrual dating or ultrasound of a natural pregnancy.
* Singleton fetus
* No evidence of abnormal nuchal thickening on preliminary ultrasound prior to chorion villus biopsy

Exclusion Criteria:

* Pregnancy by in vitro fertilization
* Evidence of a nuchal translucency of > 3.0 mm at the time of the ultrasound for the chorion villus biopsy.
* HIV, hepatitis C or hepatitis B positive maternal status
* Active infection in the mother at the time of scheduled CVS or cell injection as determined by clinical practice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
To determine whether immune tolerance and donor cell engraftment can be achieved through first trimester injection of donor cells to fetus's diagnosed with lethal LSDs. | after 3 patients
Safety and feasibility of fetal intrap. | after 3 patients

SECONDARY OUTCOMES:
Donor chimerism for neonate at birth and 7 days post delivery. | after 3 patients
Establishment of threshold enzyme levels in neonate at birth and 7 days post delivery. | after 3 patients
Donor chimerism for mother post delivery and 1 year post date of birth. | after 3 patients

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center Pediatric Blood and Marrow Transplant, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No